CLINICAL TRIAL: NCT04259697
Title: Comparison of the Effects of Clinical Pilates and Whole Body Vibration Exercises on Strength, Flexibility, Balance, Bone Turnover Markers and Quality of Life in Postmenopausal Osteoporotic Women
Brief Title: Effects of Clinical Pilates and Whole Body Vibration Exercises in Postmenopausal Osteoporotic Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Burcu Ece KORKMAZ, Principal Investigator, Dokuz Eylul University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ece Korkmaz
Record Dates: First submitted 2020-02-02; First posted 2020-02-06 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Osteoporosis
Keywords: postmenopausal osteoporosis; clinical pilates; whole body vibration; bone turnover markers; strength; flexibility; balance; quality of life
MeSH Terms: conditions — Osteoporosis; Osteoporosis, Postmenopausal

STUDY DESIGN:
Intervention Model Description: A controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinical pilates (Experimental): Exercises will be performed two times per week for twelve weeks.
  Interventions: Other: Clinical pilates
- Whole body vibration (Experimental): Exercises will be performed two times per week for twelve weeks.
  Interventions: Other: Whole body vibration

INTERVENTIONS:
Other: Clinical pilates — Clinical pilates exercises will be performed progressively. The duration of each exercise session will be an average of 40 minutes initially and then will be increased to 60 minutes as the program progress.
  Arms: Clinical pilates
Other: Whole body vibration — Whole body vibration exercises will be performed using the Power Plate pro5 AIRdaptive machine.The duration of each exercise session will be an average of 20 minutes initially and then will be increased to 30 minutes as the program progress.
  Arms: Whole body vibration

SUMMARY:
The aim is to compare the effects of clinical pilates and whole body vibration exercises in postmenopausal osteoporotic women on strength, flexibility, balance, bone turnover markers and quality of life.

DETAILED DESCRIPTION:
The aim of this study is to compare the effects of clinical pilates and whole body vibration exercises in postmenopausal osteoporotic women in terms of strength, flexibility, balance, bone turnover markers and quality of life. Thirty-four women who are diagnosed with postmenopausal osteoporosis will be recruited into the study. Participants will be divided into two groups: (1) clinical pilates group, (2) vibration exercises group. Exercise programs will be performed two times per week for twelve weeks. The strength of the extensor muscles of the hip, knee, back, elbow will be measured with a hand-held dynamometer. Flexibility will be assessed measuring the fingertip-to-floor distance in flexion and lateral bending. The balance performance will be assessed using the timed up and go test, Tetrax fall index and the maximum hold time on unipedal stance and on tandem stance. The short form-12 questionnaire will be used to assess the quality of life. Also, bone turnover markers will be measured. All assessments will be performed before and after exercise programs.

ELIGIBILITY:
Inclusion Criteria:

* Being in the postmenopausal period
* Having body mass index equal to or greater than 18,5 kg/m²
* A lack of regular exercise
* Having been diagnosed with osteoporosis
* Having the ability to walk independently

Exclusion Criteria:

* Having a cardiopulmonary problem that may prevent participating in exercise programs
* Having kidney stones
* Being diagnosed with diabetes
* Presence of epilepsy
* Having cardiological problems such as arrhythmia, using a pacemaker, hypertension
* Having neurological disorders such as Parkinson, stroke, multiple sclerosis, neuropathy
* Having surgery in the last 6 months

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2018-01-15 (Actual); Primary Completion 2020-04-15 (Estimated); Study Completion 2020-05-15 (Estimated)

PRIMARY OUTCOMES:
Strength | Change in strength measures from baseline to twelve weeks
  The strength of the extensor muscles of the hip, knee, back, elbow will be assessed with a hand-held dynamometer.
Flexibility | Change in flexibility measures from baseline to twelve weeks
  Flexibility wil be assessed measuring the fingertip-to-floor distance in flexion and lateral bending.
Timed up and go test | Change in Timed up and go test from baseline to twelve weeks
  Timed up and go test will be used to assess dynamic balance.
The maximum hold time on unipedal stance and on tandem stance. | Change in the maximum hold time from baseline to twelve weeks
  The maximum hold time will be calculated to assess static balance.
Tetrax fall index | Change in Tetrax fall index from baseline to twelve weeks
  Tetrax fall index will be calculated to determine fall risk.
The short form-12 questionnaire | Change in quality of life measure from baseline to twelve weeks
  The short form-12 questionnaire will be used to assess quality of life. The total score can range from 0 to 100. Lower SF-12 score indicated poorer physical and mental health.
Dual-energy X-ray absorptiometry of hip and lumbar spine | Change in the Dual-energy X-ray absorptiometry of hip and lumbar spine from baseline to twelve weeks
  Dual-energy X-ray absorptiometry of hip and lumbar spine will be measured to assess bone density.
Plasma sclerostin concentration | Change in plasma sclerostin concentration from baseline to twelve weeks
  Plasma sclerostin concentration will be measured to assess the process of bone resorption and formation.
Urinary deoxypyridinoline | Change in urinary deoxypyridinoline level from baseline to twelve weeks
  Urinary deoxypyridinoline level will be measured to assess bone resorption.

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylul University, School of Physical Therapy and Rehabilitation, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided